CLINICAL TRIAL: NCT00785824
Title: A Prospective Cohort Pilot Study of Bone Metabolism in Lactating and Non-lactating Postpartum African-American Women and Healthy Non-pregnant African-American Women
Brief Title: African-American Bone Metabolism and Lactation Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mara Horwitz, Associate Professor of Medicne, University of Pittsburgh
Other Study IDs: PRO08080129; R01DK073039 (NIH)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Lactation; Bone Diseases, Endocrine
Keywords: Lactation; Endocrine System Diseases; Musculoskeletal System Disease; Hormone; Physiological Properties
MeSH Terms: conditions — Breast Feeding; Bone Diseases, Endocrine; Endocrine System Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — archival blood serum and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1 A-A Breastfeeding Mothers: Group 1: Postpartum African-American breastfeeding women at 6-8 weeks post childbirth, and again at 12-14 weeks post childbirth
- 2 - AA Bottlefeeding Mothers: Group 2: Postpartum African-American bottlefeeding women at 6-8 weeks post childbirth and again at 12-14 weeks post childbirth.
- 3 - AA Normal Controls: Group 3: Normal African-American non-pregnant controls who are age-matched to Group 1

SUMMARY:
The primary aim of this study is to obtain measures of amino-terminal telopeptides of procollagen 1 (P1NP), a marker of bone formation, in lactating and non-lactating post-partum African-American women both at 6-8 and at 12-14 weeks post-partum, and to compare these values to those of normal controls. The secondary aim is to obtain at the same time points, measurements of Parathyroid Hormone-related Protein (PTHrP), additional markers of bone turnover [e.g. N-telopeptide of collagen cross-links (NTx), C-telopeptide of collagen cross-links (Ctx),bone specific alkaline phosphatase (BSAP) and osteocalcin (OC)], calcium and vitamin D metabolism in these subjects. These results will be compared with a non-African-American cohort of post-partum women and normal controls.

The investigators hypothesize that African-American lactating women will have increased bone turnover when compared to non-lactating postpartum women and normal controls. The investigators further hypothesize that bone turnover is increased in lactating women independent of race.

DETAILED DESCRIPTION:
Pregnancy and lactation are both states of altered maternal calcium and bone metabolism which may have a significant impact on the development of peak bone mass. While these two states are characterized by different hormonal environments, both have been associated with significant bone loss. The maternal hormonal mechanism for providing calcium to meet the needs of the developing fetus appear different from those that meet the needs of lactation. During pregnancy, the 30 gm of calcium required by the fetus comes predominantly from an increase in maternal intestinal calcium absorption which is mediated by 1,25 dihydroxy vitamin D and other factors. Several studies have measured total and free 1,25 dihydroxy vitamin D through pregnancy and find the values nearly double. Serum Parathyroid Hormone (PTH) levels fall to about 10-30% of the mean non-pregnant value in the first trimester and then increase to the mid-normal range by term, while ionized calcium remains normal throughout pregnancy. Parathyroid Hormone-related Protein (PTHrP) levels gradually increase throughout pregnancy although the source (maternal, fetal, or placental) remains unclear. Most studies of bone metabolism in humans during pregnancy have measured changes in markers of bone turnover rather than bone density to avoid radiation exposure to the fetus. These studies have been confounded by several variables such as the effects of hemodilution in pregnancy, altered glomerular filtration rates (GFR), degradation and clearance of markers by the placenta, which may cloud the results. Some of these studies report an increase in urinary markers of bone resorption from early to mid pregnancy while bone formation markers decrease and then rise before term. Importantly, no one has assessed state-of-the-art markers of bone formation such as type 1 Procollagen N-terminal Propeptide (P1NP) in pregnancy or lactation.

During lactation in humans, it is estimated that 600 to 1000 ml of milk are produced a day with daily calcium loss of 200 to 400 mg. In contrast to pregnancy, a majority of this calcium comes from demineralization of the maternal skeleton, and is probably predominately mediated by PTHrP in the setting of low estrogen. PTHrP levels are significantly higher in lactating women than non-lactating controls while intact PTH is reduced by approximately 50% during the first several months of lactation. The source of the PTHrP is likely the mammary gland, as PTHrP levels are elevated 10,000 fold in milk and circulating maternal PTHrP levels are increased further with suckling. This is also supported by a mouse model in which the tissue-specific ablation of the PTHrP gene in the lactating mammary gland resulted is a decrease in bone loss during lactation. When PTHrP enters the maternal circulation, it stimulates maternal bone resorption from the skeleton and renal tubular resorption of calcium. PTHrP indirectly suppresses PTH as ionized calcium rises to upper levels of normal. 1,25 dihydroxyvitamin D levels fall to within the normal range during lactation, although they have been reported to be higher in lactating than non-lactating postpartum women. Intestinal absorption of calcium also returns to normal during the post-partum period. Serial bone density measurement (BMD)obtained during lactation show a fall of 3-10% in trabecular bone (spine, hip, femur) with a smaller 1-2% loss at cortical bone. Both losses are far greater that than that seen in early postmenopausal women, or in women receiving gonadotropin releasing hormone (GnRH) agonist therapy. This implies that it is not only the fall in estrogen that mediates bone loss during lactation. The bone loss during lactation seems to be transient as there is rapid recovery of bone density in postpartum women with weaning and the resumption of menses.

Markers of bone resorption have been measured in urine in several prospective studies of lactation in humans where they have been reported to be elevated 2-3 fold. However, these results may be confounded by a decrease in GFR and volume contraction that may occur during lactation compared to pregnancy. Surprisingly, more reliable markers of bone resorption measured in serum (CTX and NTX) have not been measured in a controlled lactation study. Markers of bone formation as measured by osteocalcin (Oc) and bone specific alkaline phosphatase (BSAP) have generally been reported to be higher during lactation. However, these results are difficult to interpret as BSAP is not a very sensitive marker of bone formation. Recent data has emerged suggesting that Oc may measure bone resorption as well as formation. The current most accurate measure of bone formation is serum amino-terminal telopeptides of procollagen 1 (P1NP), which until recently had not been measured in a control study of lactating women. We are currently analyzing data from a controlled study of lactation in Caucasian, Hispanic, and Asian women.

Most of the studies on bone metabolism during pregnancy and lactation have been performed in Caucasian females. Most studies have excluded African-Americans due to the unique differences in bone metabolism known to occur in this population which may create wider statistical variation in the study results.

It is well established that bone metabolism in African American subjects differs from the Caucasians in several aspects. The mean 25-hydroxyvitamin D levels are lower in African-Americans primarily due to reduced vitamin D production in the skin associated with increased pigmentation as well as reduced intake of vitamin D. As a consequence, African-Americans have relative secondary hyperparathyroidism and resultant higher levels of PTH, and 1, 25 dihydroxyvitamin D, and lower urinary calcium excretion. One would expect that patients with secondary hyperparathyroidism would result in increased bone turnover and decreased bone mass. This is not what is observed in African Americans though. African Americans have higher bone density and lower fracture risk as compared to Caucasians. Moreover, biochemical markers of bone turnover in African-Americans are in general lower than in Caucasians, particularly for bone formation, as measured by osteocalcin. On the other hand, there is normal or increased renal absorption of calcium. Based on these, Dr. Normal Bell proposed that the black skeleton is resistant to the effects of PTH, while renal sensitivity is maintained or even enhanced. This hypothesis is further supported by the observation of significantly lower bone resorption (as measured by cross-linked N-telopeptide of procollagen I (NTx), cross-linked C-telopeptide of type I collagen (CTx), and free deoxypyridinoline (DPD) and normal to low renal excretion of calcium in response to PTH infusion in African American as compared with Caucasian women.

This is a prospective cohort study of post-partum lactating, non-lactating, and healthy control African-American women who are not currently or have not recently been pregnant. The investigators hope to estimate the measurable differences in bone formation and resorption by comparing blood and urine samples from African-American lactating women to African-American non-lactating postpartum women and normal controls. 100 female volunteers between the ages of 21-45 years will be recruited to achieve 75 evaluable subjects or 25 in each of the three groups. There are two out-patient visits, each 6-8 weeks apart. The visits will take place at the University of Pittsburgh Medical Center (UPMC) - Clinical & Translational Research Center (CTRC) located on 6 North East (6 NE) in Montefiore Hospital. The post-partum subjects will be recruited during their last trimester of pregnancy or at their 6-week post-partum visit. Healthy controls will be recruited and matched to a breast-feeding postpartum woman who has already completed the study. Visit 1 for all postpartum women will take place at 6-8 weeks after delivery and Visit 2 at 14 weeks after delivery. Healthy control subjects will have two study visits at similar intervals to their matched breast-feeding subject (1.5 to 2 months). For all subjects, an informed consent will be obtained at the first visit, before any study procedures are done: including a medical history and measurement of vital signs, an intake history about menstrual cycles, pregnancy, and if applicable, delivery and breast or bottle feeding events. Subjects will complete a dietary calcium intake questionnaire. Blood collections are obtained at each visit for measurements of the following: serum ionized and total calcium, phosphorus, creatinine, albumin, PTH(1-34), PTH(1-84), PTHrP (1-36), 25-hydroxy Vitamin D by High Performance Liquid Chromatography (HPLC), including D2 and D3, 1,25 (OH)2 vitamin D, estrogen status, Luteinizing Hormone (LH), Follicle-stimulating Hormone (FSH), Estradiol, and markers of bone metabolism (e.g. NTX, CTX, P1NP, Osteocalcin (OC), BSAP, Insulin-like growth factor-1 (IGF-1), and selected cytokines of the interleukin-6 (IL-6). Urine samples will be obtained for calcium, creatinine and phosphorus. A urine pregnancy test will be done at each visit for normal controls. Post-partum women will have a urine pregnancy checked at Visit 2 only, to avoid false positives that are likely at Visit 1 due to the recently completed pregnancy. Thyroid Stimulating Hormone (TSH) will be checked at Visit 1 to exclude those women who have significant alterations in thyroid functioning that could interfere with bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Post-partum (singleton pregnancy) African-American women who are exclusively breastfeeding, defined as 1 or fewer bottles of supplemental formula/day.
* Group 2: Post-partum (singleton pregnancy) African-American women are non-lactating, which is defined as bottle-feeding or having weaned their baby from breastfeeding for at least 4 weeks prior to study.
* Group 3: Controls- Healthy non-pregnant African-American women will be race and age-matched to the breast-feeding women in group one. They may not have been lactating or pregnant within the last year.

Exclusion Criteria:

* Subjects with cardiac, hypertensive, vascular, renal (serum creatinine of >1.5), pulmonary, endocrine, musculoskeletal, hepatic, hematologic or malignant or rheumatologic disease will be excluded from the study.
* Smokers and those with a history of significant alcohol or drug abuse are excluded.
* Baseline hypertension (systolic BP > 160 mm/Hg) or hypotension (systolic BP < 90 mm/Hg).
* Subjects taking any chronic medications except stable doses of thyroid hormone, prenatal, vitamin supplements, or oral contraceptives.
* Those who have received any investigational drug in past 90 days will be excluded from the study.
* Women who are currently pregnant will be excluded from the study. Women who became pregnant by In Vitro Fertilization IVF or any hormonal manipulation (i.e. fertility drugs such as clomid ®) are also excluded, as they may have an altered pre-pregnant hormonal state. All women will have a urine pregnancy test performed at each of the two study visits and must not be pregnant in order to continue in the study. Subjects are not allowed to donate blood between study visits.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: New African-American mothers who are either almost exclusively breast-feeding or bottle-feeding; normal controls to match the lactating mothers
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Measurements of amino-terminal telopeptides of procollagen 1 (P1NP), a marker of bone formation, in lactating and non-lactating post-partum African-American women both at 6-8 and at 12-14 weeks post-partum and normal controls | 4 months

SECONDARY OUTCOMES:
Measurements of Parathyroid Hormone-related Protein (PTHrP), additional markers of bone turnover (i.e. NTX - N-telopepetide of collagen cross-links, CTX - C-telopepetide of collagen cross-links, BSAP - bone specific alkaline phosphatase and osteocalcin), | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mara J Horwitz, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Dobnig H, Kainer F, Stepan V, Winter R, Lipp R, Schaffer M, Kahr A, Nocnik S, Patterer G, Leb G. Elevated parathyroid hormone-related peptide levels after human gestation: relationship to changes in bone and mineral metabolism. J Clin Endocrinol Metab. 1995 Dec;80(12):3699-707. doi: 10.1210/jcem.80.12.8530622.
- [Background] Gundberg CM, Looker AC, Nieman SD, Calvo MS. Patterns of osteocalcin and bone specific alkaline phosphatase by age, gender, and race or ethnicity. Bone. 2002 Dec;31(6):703-8. doi: 10.1016/s8756-3282(02)00902-x. PMID 12531565
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Hollis BW, Garcia-Ocana A, Stewart AF. Direct comparison of sustained infusion of human parathyroid hormone-related protein-(1-36) [hPTHrP-(1-36)] versus hPTH-(1-34) on serum calcium, plasma 1,25-dihydroxyvitamin D concentrations, and fractional calcium excretion in healthy human volunteers. J Clin Endocrinol Metab. 2003 Apr;88(4):1603-9. doi: 10.1210/jc.2002-020773. PMID 12679445
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Syed MA, Garcia-Ocana A, Bisello A, Hollis BW, Rosen CJ, Wysolmerski JJ, Dann P, Gundberg C, Stewart AF. Continuous PTH and PTHrP infusion causes suppression of bone formation and discordant effects on 1,25(OH)2 vitamin D. J Bone Miner Res. 2005 Oct;20(10):1792-803. doi: 10.1359/JBMR.050602. Epub 2005 Jun 6. PMID 16160737
- [Background] Kalkwarf HJ, Specker BL, Ho M. Effects of calcium supplementation on calcium homeostasis and bone turnover in lactating women. J Clin Endocrinol Metab. 1999 Feb;84(2):464-70. doi: 10.1210/jcem.84.2.5451. PMID 10022402
- [Background] Kovacs CS. Calcium and bone metabolism during pregnancy and lactation. J Mammary Gland Biol Neoplasia. 2005 Apr;10(2):105-18. doi: 10.1007/s10911-005-5394-0. PMID 16025218
- [Background] Kovacs CS, Kronenberg HM. Maternal-fetal calcium and bone metabolism during pregnancy, puerperium, and lactation. Endocr Rev. 1997 Dec;18(6):832-72. doi: 10.1210/edrv.18.6.0319. No abstract available. PMID 9408745
- [Background] Sowers M, Eyre D, Hollis BW, Randolph JF, Shapiro B, Jannausch ML, Crutchfield M. Biochemical markers of bone turnover in lactating and nonlactating postpartum women. J Clin Endocrinol Metab. 1995 Jul;80(7):2210-6. doi: 10.1210/jcem.80.7.7608281.
- [Background] Sowers MF, Hollis BW, Shapiro B, Randolph J, Janney CA, Zhang D, Schork A, Crutchfield M, Stanczyk F, Russell-Aulet M. Elevated parathyroid hormone-related peptide associated with lactation and bone density loss. JAMA. 1996 Aug 21;276(7):549-54. PMID 8709404
- [Background] VanHouten JN, Dann P, Stewart AF, Watson CJ, Pollak M, Karaplis AC, Wysolmerski JJ. Mammary-specific deletion of parathyroid hormone-related protein preserves bone mass during lactation. J Clin Invest. 2003 Nov;112(9):1429-36. doi: 10.1172/JCI19504. PMID 14597768
- [Background] Bell NH, Yergey AL, Vieira NE, Oexmann MJ, Shary JR. Demonstration of a difference in urinary calcium, not calcium absorption, in black and white adolescents. J Bone Miner Res. 1993 Sep;8(9):1111-5. doi: 10.1002/jbmr.5650080912. PMID 8237481
- [Background] Cosman F, Morgan DC, Nieves JW, Shen V, Luckey MM, Dempster DW, Lindsay R, Parisien M. Resistance to bone resorbing effects of PTH in black women. J Bone Miner Res. 1997 Jun;12(6):958-66. doi: 10.1359/jbmr.1997.12.6.958. PMID 9169356
- [Background] Finkelstein JS, Lee ML, Sowers M, Ettinger B, Neer RM, Kelsey JL, Cauley JA, Huang MH, Greendale GA. Ethnic variation in bone density in premenopausal and early perimenopausal women: effects of anthropometric and lifestyle factors. J Clin Endocrinol Metab. 2002 Jul;87(7):3057-67. doi: 10.1210/jcem.87.7.8654. PMID 12107201
- [Background] Fuleihan GE, Gundberg CM, Gleason R, Brown EM, Stromski ME, Grant FD, Conlin PR. Racial differences in parathyroid hormone dynamics. J Clin Endocrinol Metab. 1994 Dec;79(6):1642-7. doi: 10.1210/jcem.79.6.7989469.
- [Background] George A, Tracy JK, Meyer WA, Flores RH, Wilson PD, Hochberg MC. Racial differences in bone mineral density in older men. J Bone Miner Res. 2003 Dec;18(12):2238-44. doi: 10.1359/jbmr.2003.18.12.2238. PMID 14672360
- [Background] Perry HM 3rd, Horowitz M, Morley JE, Fleming S, Jensen J, Caccione P, Miller DK, Kaiser FE, Sundarum M. Aging and bone metabolism in African American and Caucasian women. J Clin Endocrinol Metab. 1996 Mar;81(3):1108-17. doi: 10.1210/jcem.81.3.8772584.
- [Background] Nelson DA, Barondess DA, Hendrix SL, Beck TJ. Cross-sectional geometry, bone strength, and bone mass in the proximal femur in black and white postmenopausal women. J Bone Miner Res. 2000 Oct;15(10):1992-7. doi: 10.1359/jbmr.2000.15.10.1992. PMID 11028452
- [Background] Carneiro RM, Prebehalla L, Tedesco MB, Sereika SM, Hugo M, Hollis BW, Gundberg CM, Stewart AF, Horwitz MJ. Lactation and bone turnover: a conundrum of marked bone loss in the setting of coupled bone turnover. J Clin Endocrinol Metab. 2010 Apr;95(4):1767-76. doi: 10.1210/jc.2009-1518. Epub 2010 Feb 11. PMID 20150580
- [Derived] Carneiro RM, Prebehalla L, Tedesco MB, Sereika SM, Gundberg CM, Stewart AF, Horwitz MJ. Evaluation of markers of bone turnover during lactation in African-Americans: a comparison with Caucasian lactation. J Clin Endocrinol Metab. 2013 Feb;98(2):523-32. doi: 10.1210/jc.2012-2118. Epub 2012 Dec 28. PMID 23275526